CLINICAL TRIAL: NCT05596266
Title: A Phase I Study of CD5 CAR-T for Refractory/Relapsed CD5+ T-ALL Patients
Brief Title: CD5 CAR-T Therapy for Refractory/Relapsed CD5+ T-cell Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Baoding Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202001
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: T-cell Acute Lymphoblastic Leukemia
Keywords: CD5 CAR-T; T-ALL
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD5 CAR-T (Experimental): This cohort will be administrated with T cells transduced with lentivirus vectors expressing CD5 CAR.
  Interventions: Biological: CD5 CAR-T

INTERVENTIONS:
Biological: CD5 CAR-T — CD5 CAR-T will be administered by I.V. infusion.

SUMMARY:
This is a phase I, interventional, single arm, open label, clinical study to evaluate the safety and tolerability of CD5 CAR-T cells in refractory/relapsed CD5+ T-ALL patients who have no available curative treatment options.

DETAILED DESCRIPTION:
T-acute lymphoblast leukemia (T-ALL) is a neoplastic lymphoid leukemia characterized by the proliferation of immature precursor T cells. The combined chemotherapy has significantly improved the prognosis of T-acute lymphoblast leukemia/lymphoma. However, once the disease appears to be relapsed/refractory, there is limited treatment options, and the overall prognosis is extremely poor. Therefore, exploring safe and effective treatments is a critical unmet medical need. The patients will receive infusion of CAR T-cells targeting CD5 to examine the safety and, possibly the efficacy of CD5 CAR T-Cells in CD5+ relapsed or refractory acute leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of refractory or relapsed T-cell acute lymphoblastic leukemia (T-ALL) according to the NCCN 2019.V2 Guideline. Refractory T-ALL is defined as a patient who has failed to achieve complete remission after induction therapy. Relapsed T-ALL is defined as the reappearance of blasts (5%) in either peripheral blood or bone marrow. Patients whose tumor burden >5% blasts, or who have persistent positive minimal residual disease (MRD), or have reappearance of extramedullary lesions are also considered eligible;
2. CD5-positive tumor (≥70% CD5 positive blasts by flow cytometry or immunohistochemistry (tissue) assessed by a CLIA certified Flow Cytometry/Pathology laboratory). tumors burden >5%,or MRD+， or new extramedullary lesions reappeared;
3. Aged 1 to 18 years (including 18 years old);
4. Eastern Cooperative Oncology Group (ECOG) score 0-2;
5. Life expectancy greater than 12 weeks;
6. Oxygen saturation of blood>90%;
7. Total bilirubin (TBil) ≤3 × upper limit normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 10 × upper limit of normal;
8. Informed consent explained to, understood by and signed by patient/guardian.

Exclusion Criteria:

1. Intracranial hypertension or brain consciousness disorder;
2. Has an active GvHD;
3. Has a history of severe pulmonary function damaging;
4. With other tumors which is/are in advanced malignant stage and has/have systemic metastasis;
5. Severe or persistent infection that cannot be effectively controlled；
6. Presence of severe autoimmune diseases or immunodeficiency disease;
7. Patients with active hepatitis B or hepatitis C ([HBVDNA+] or [HCVRNA+]);
8. Patients with HIV infection or syphilis infection;
9. Has a history of serious allergies to biological products (including antibiotics);
10. Clinically significant viral infection or uncontrolled viral reactivation of EBV (Epstein-Barr virus), CMV (cytomegalovirus), ADV (adenovirus), BK-virus, or HHV (human herpesvirus)-6;
11. Presence of any symptomatic CNS disorder such as an uncontrolled seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement;
12. Received allogeneic hematopoietic stem cell transplantation within 6 months;
13. Being pregnant and lactating or having pregnancy within 12 months;
14. Any situations that the researchers believe will increase the risk for the subject or affect the results of the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-25 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 1 month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within the first one month following CD5 CAR-T infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity.

SECONDARY OUTCOMES:
Efficacy: Remission Rate | 1 months post CAR-T cells infusion
  Remission Rate including complete remission(CR)、CR with incomplete blood count recovery(CRi)、partial remission(PR), No remission(NR), overall remission (OR).
Best overall response (BOR) | 1 months
  Best overall response (BOR) of complete remission (CR) or CR with incomplete blood count recovery (CRi) within 1 months after CD5 CAR-T infusion.
Duration of remission (DoR) | 1 year
  Duration of remission (DoR) within 1 year following CD5 CAR-T infusion (DoR is defined as the duration from the date when the response criteria of CR or CRi is first met to the date of relapse or death due to ALL).
Event free survival within 1 year | 1 year
  Event free survival (EFS) within 1 year (EFS is defined as the time from start of the first infusion to the earliest of death from any cause or relapse).

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Chen, PhD, Principal Investigator — Xuanwu Hospital, Beijing; Huyong Zheng, MD, PhD, Principal Investigator — Baoding Children's Hospital; Beijing Children's Hospital, Capital Medical University
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China